CLINICAL TRIAL: NCT01699750
Title: Comparative In-Vivo Wetting Characteristics of Silicone Hydrogel Materials With Selected Lens Care Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: M-12-043 / ID11-59
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Myopia; Astigmatism; Refractive Error
Keywords: contact lenses; contact lens solution; myopia; astigmatism
MeSH Terms: conditions — Myopia; Astigmatism; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Air Optix Aqua (Experimental): Lotrafilcon B contact lenses with OFPM and BIOTRUE for 30 days each
  Interventions: Device: Lotrafilcon B contact lenses; Device: OPTI-FREE® PUREMOIST® MPDS; Device: BIOTRUE®; Device: Balafilcon A contact lenses; Device: ReNu® Multiplus®
- Acuvue Oasys (Active Comparator): Senofilcon A contact lenses with OFPM and BIOTRUE for 30 days each
  Interventions: Device: Senofilcon A contact lenses; Device: OPTI-FREE® PUREMOIST® MPDS; Device: BIOTRUE®; Device: Balafilcon A contact lenses; Device: ReNu® Multiplus®

INTERVENTIONS:
Device: Lotrafilcon B contact lenses — Silicone hydrogel contact lenses, Phase 2
  Other Names: AIR OPTIX® AQUA; AOA
  Arms: Air Optix Aqua
Device: Senofilcon A contact lenses — Silicone hydrogel contact lenses, Phase 2
  Other Names: ACUVUE® OASYS® with HYDRACLEAR®; AVO
  Arms: Acuvue Oasys
Device: OPTI-FREE® PUREMOIST® MPDS — Contact lens care system, Phase 2
  Other Names: OFPM
Device: BIOTRUE® — Contact lens care system, Phase 2
Device: Balafilcon A contact lenses — Silicone hydrogel contact lenses worn for 30 days, Phase 1
  Other Names: PureVision
Device: ReNu® Multiplus® — Contact lens care system used for 30 days, Phase 1

SUMMARY:
The purpose of this study is to evaluate the lipid uptake, wetting characteristics, and visual performance of AIR OPTIX® AQUA and ACUVUE® OASYS® with HYDRACLEAR® contact lenses when used in conjunction with two contact lens care systems.

DETAILED DESCRIPTION:
This study will be divided into two phases. In the Pre-Investigational Phase (Phase 1), participants will wear PureVision contact lenses for 30 days and use ReNu® Multiplus® for contact lens care. Eligible participants will continue into the Investigational Phase (Phase 2) and be randomly assigned to wear AIR OPTIX® AQUA contact lenses or ACUVUE® OASYS® with HYDRACLEAR® contact lenses for a total of two months. For contact lens care, participants will use OPTI-FREE® PUREMOIST® MPDS and BIOTRUE® for 30 days each.

ELIGIBILITY:
Inclusion Criteria:

* Read and understand the Participant Information Sheet;
* Read, sign, and date the Informed Consent;
* Be a current silicone hydrogel contact lens wearer using the contact lenses under a frequent replacement (bi-weekly or monthly) daily wear modality;
* Be classified as symptomatic and a depositor at the end of the replacement period according to protocol-specified criteria;
* Agree to wear study contact lenses as directed for the duration of the study and maintain the appointment schedule;
* Best corrected visual acuity of 6/9 or better in each eye;
* Normal eyes with the exception of the need for visual correction;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known sensitivity or intolerance to any of the contact lenses or contact lens care products to be used;
* Monocular vision (only one eye with functional vision or only one eye fitted with contact lenses);
* Use of systemic medication which might interfere with contact lens wear or produce dry eye side effects;
* Systemic disease which might interfere with contact lens wear or produce dry eye side effects;
* Systemic or ocular allergies which might interfere with contact lens wear;
* Ocular disease which might interfere with contact lens wear;
* Active ocular infection;
* Use of any concomitant topical ocular medications during the study period;
* Previous ocular surgery;
* Pregnant, planning to become pregnant, or lactating at the time of enrollment;
* Participation in an investigational drug or device study within 30 days of entering this study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kern, PhD, Study Director — Alcon Research
Locations (1):
- Contact Alcon Call Center at 1-888-451-3937 for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in the United Kingdom.
Pre-assignment Details: Of the 109 participants enrolled, 39 were exited from the study prior to randomization and product dispense (Phase 2). This reporting group includes all randomized and dispensed participants (70).
Period: Overall Study
Arm/Group | Air Optix Aqua | Acuvue Oasys
Started | 34 | 36
Completed | 34 | 33
Not Completed | 0 | 3
Not completed — Withdrew Consent | 0 | 1
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized and dispensed participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Air Optix Aqua | Acuvue Oasys | Total
Number analyzed (Participants) | 34 | 36 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (10.95) | 35.3 (8.77) | 35.6 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 10 | 7 | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Ex-Vivo Total Lipid Uptake Per Lens
Description: The contact lens was aseptically removed from the eye. Lipids were extracted and analyzed using a proprietary High Performance Liquid Chromatography technique. A lower value indicates a cleaner lens surface. One eye (study eye) contributed to the mean.
Time Frame: Day 30
Population: This analysis group includes all participants who had a baseline and at least one post-baseline measurement of the primary efficacy endpoint. Two Day 30 measurements per participant (one eye per Day 30) contributed to analysis.
Measure: Geometric Mean (Standard Deviation); unit: micrograms
Arm/Group | Air Optix Aqua | Acuvue Oasys
Number analyzed (Participants) | 34 | 33
micrograms | 7.198 (1.5014) | 35.879 (1.8185)

2. Secondary Outcome: Mean Non-Invasive Pre-Lens Tear Film Break Up Time (NIBUT)
Description: The pre-lens tear film is the layer of tears located on top of the contact lens between the eyelid and the contact lens. NIBUT (i.e., the time elapsed between eye opening after a blink and the appearance of the first dark spot within the tear film) was measured using a diffuse illumination source (Tearscope) and videotography. A longer NIBUT indicates a more stable tear film and greater on-eye lens wettability. One eye (study eye) contributed to the mean.
Time Frame: Day 30
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: seconds
Arm/Group | Air Optix Aqua | Acuvue Oasys
Number analyzed (Participants) | 34 | 33
seconds | 3.316 (2.6913) | 2.918 (2.4859)

3. Secondary Outcome: LogMAR Time-Controlled Visual Acuity (TCVA)
Description: Visual performance was measured binocularly (both eyes together) at two contrast levels using a validated Time Controlled Visual Acuity test (TCVA). TCVA was recorded in VA units (1 VA unit=1 VA line=0.1 logMAR), with positive (+) values corresponding with VA better than 20/20 and negative (-) values worse than 20/20.
Time Frame: Day 30
Population: This analysis group includes all participants who had a baseline and at least one post-baseline measurement of the primary efficacy. Two Day 30 measurements per participant contributed to analysis.
Measure: Mean (Standard Deviation); unit: VA unit
Arm/Group | Air Optix Aqua | Acuvue Oasys
Number analyzed (Participants) | 34 | 33
VA unit
  High Contrast | 0.38 (1.058) | -0.14 (0.999)
  Low Contrast | -1.15 (1.213) | -1.60 (1.040)

4. Secondary Outcome: Overall Comfort Measured With Visual Analog Scale (VAS)
Description: The participant rated overall comfort on a 100-millimeter analog scale by marking a line that best corresponds to their eye comfort (0=very poor, 100=excellent). Both eyes were rated together as a single, retrospective evaluation of the previous 3 days of wear.
Time Frame: Day 30
Population: This analysis group includes all participants who had a baseline and at least one post-baseline measurement of the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- OFPM With Air Optix Aqua: OFPM with lotrafilcon B contact lenses for 30 days
- OFPM With Acuvue Oasys: OFPM with senofilcon A contact lenses for 30 days
- BIOTRUE With Air Optix Aqua: BIOTRUE with lotrafilcon B contact lenses for 30 days
- BIOTRUE With Acuvue Oasys: BIOTRUE with senofilcon A contact lenses for 30 days
Arm/Group | OFPM With Air Optix Aqua | OFPM With Acuvue Oasys | BIOTRUE With Air Optix Aqua | BIOTRUE With Acuvue Oasys
Number analyzed (Participants) | 34 | 33 | 34 | 33
units on a scale | 77.1 (20.25) | 81.1 (20.37) | 74.9 (28.43) | 82.2 (20.76)

5. Secondary Outcome: Overall Dryness Measured With Visual Analog Scale (VAS)
Description: The participant rated overall dryness on a 100-millimeter analog scale by marking a line that best describes how dry their eyes feel (0=not at all dry, 100=very dry). Both eyes were rated together as a single, retrospective evaluation of the previous 3 days of wear.
Time Frame: Day 30
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OFPM With Air Optix Aqua | OFPM With Acuvue Oasys | BIOTRUE With Air Optix Aqua | BIOTRUE With Acuvue Oasys
Number analyzed (Participants) | 34 | 33 | 34 | 33
units on a scale | 21.8 (20.41) | 22.2 (22.15) | 23.3 (25.65) | 22.5 (25.60)

6. Secondary Outcome: Average Exposure Speed
Description: Exposure speed (rate of increase in exposed lens surface % (areas not protected by tear film) after the first tear film break and before the second blink) was measured with a diffuse illumination source (Tearscope) and videotography. Higher speeds indicate worse tear film dynamics. One eye (study eye) contributed to the mean.
Time Frame: Day 30
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: percent of area exposed/second
Arm/Group | Air Optix Aqua | Acuvue Oasys
Number analyzed (Participants) | 34 | 33
percent of area exposed/second | 0.059 (15.1175) | 0.105 (24.4808)

7. Secondary Outcome: Minimum Protected Area
Description: Minimum protected area (i.e., minimum area of the lens (%) covered by the tear film during the interblink period) was measured using a diffuse illumination source (Tearscope) and videotography. A higher value indicates a larger area of the tearfilm spread evenly over the lens (i.e., less area of tear film breakage). One eye (study eye) contributed to the mean.
Time Frame: Day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of lens surface covered
Arm/Group | Air Optix Aqua | Acuvue Oasys
Number analyzed (Participants) | 34 | 33
percentage of lens surface covered | 90.75 (15.990) | 77.79 (31.547)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (December 2012-November 2013).This analysis group includes all participants randomized into the Investigational Phase of the study who participated in at least one period of the study.
Description: An adverse event was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device.
Groups:
- AIR OPTIX AQUA: Lotrafilcon B contact lenses worn for 60 days, replaced monthly
- ACUVUE OASYS With HYDRACLEAR: Senofilcon A contact lenses worn for 60 days, replaced biweekly
Arm/Group | AIR OPTIX AQUA | ACUVUE OASYS With HYDRACLEAR
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 3/34 | 7/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIR OPTIX AQUA (N=34) | ACUVUE OASYS With HYDRACLEAR (N=36)
Nasopharyngitis (Infections and infestations) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Eye complication associated with device (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.